CLINICAL TRIAL: NCT05073770
Title: A Clinical Feasibility Study to Assess the Performance of a Latex Condom in Healthy Monogamous Couples.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Titan Condoms, LLC (Industry)
Collaborators: STATCure Consulting Services Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 9289
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Performance of a New Condom

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N64 (Experimental): Based on the penis girth measurements, eligible participants will be assigned to two groups:
  Group 1: The couples who will test the 64 mm plain condom (n=25).
  The test condom has the following specifications throughout the study:
  The plain 64mm condom (i.e., N64): Length 223 ±5mm, width 64±1mm, thickness (single wall) 0.070± 0.005mm, and beading thickness 1.25±0.05mm.
  Interventions: Device: Titan Condom
- N69 (Experimental): Based on the penis girth measurements, eligible participants will be assigned to two groups:
  Group 2: The couples who will test the 69 mm plain condom (n=25).
  The test condom has the following specifications throughout the study:
  The plain 69mm condom (i.e., N69): Length 223 ±5mm, Width 69±1mm, Thickness (single wall) 0.070± 0.005mm, Beading thickness 1.25±0.05mm.
  Interventions: Device: Titan Condom

INTERVENTIONS:
Device: Titan Condom — The test condoms have the following specifications throughout the study:
  1. The plain 64mm condom (i.e., N64): Length 223 ±5mm, width 64±1mm, thickness (single wall) 0.070± 0.005mm, and beading thickness 1.25±0.05mm.
  2. The plain 69mm condom (i.e., N69): Length 223 ±5mm, Width 69±1mm, Thickness (single wall) 0.070± 0.005mm, Beading thickness 1.25±0.05mm.

SUMMARY:
The U.S. Centers for Disease Control and Prevention has recommended the male latex condom as the best physical barrier for preventing HIV and sexually transmitted disease (STD) transmission. Condoms are a safe and effective form of contraception that have 98% effectiveness in protecting against STD and pregnancy. However, evidence shows that if a condom does not fit properly, its impact can reduce to 85% or less, as it may slip off during sex or during removal of the penis from the vagina or breaks during intercourse.

Condoms need to fit correctly to guard against fluids and exposed skin which could lead to STD contraction or pregnancy. To choose the right size, the girth (the width of an erect penis) is the most important factor, not length. However, most condom companies do not list their nominal width, let alone base their sizes off girth. In addition, most brands usually offer XL as only 56 mm based on a misconception that one size fits all and that "XL" condoms are big enough. But that is far from the truth, and several men complain about the lack of simplicity and intuitiveness when finding a condom that fits them.

To address this gap, after a long two years of development, Titan company was able to engineer four distinct sizes so that each man can easily find the condom he needs. This study aims to obtain a preliminary estimate of slippage and breakage of Titan's new condom (64mm or 69mm) during use.

ELIGIBILITY:
Inclusion Criteria:

* Couples not at risk of pregnancy (using alternate contraception).
* Couples who are past or recent/experienced condom users
* No known sexually transmitted infections, including HIV/AIDS, gonorrhea, chlamydia, etc.
* Subjects between 18 to 45 years of age.
* Monogamous heterosexual couples who agree to practice vaginal sex only during the study.
* The Titan Size Guide will be used to determine subject eligibility based on the following penis girth measurements

  * Penis girth N64 ≥ 5.8"
  * Penis girth N69 ≥ 6.1"

Exclusion Criteria:

* Couples who work for the clinical testing laboratory or who are relatives of staff of the clinical test laboratory or a sponsor of the study.
* Participants with known allergy to natural rubber latex or material(s) of test condom.
* Participants with known sensitivity to the residual chemicals used in the manufacturing of natural rubber latex condoms.
* Couples where one knowingly has a sexually transmitted infection.
* Male partners have known erectile or ejaculatory dysfunction.
* Commercial sex workers.
* Female partner is pregnant or desires to become so while participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Performance (clinical slippage rate) | two-weeks
  Clinical slippage rate will be calculated as the number of condoms with at least 1 clinical slippage event divided by the number of condoms used during intercourse, reported as a percentage. Clinical slippage events, defined in ISO 29943-1:2017, will be reported by subjects. A clinical slippage is defined as a condom slipping off completely during intercourse or during withdrawal from the vagina. Slippage that occurs because the user failed to hold onto the condom at the base of the penis during withdrawal and/ or because the user delayed withdrawal after sex are to be record as "non-clinical slippage", these events are considered user failures.
Performance (clinical breakage rate) | two-weeks
  Clinical failure rate is calculated as the number of condoms with at least 1 acute clinical failure event (clinical slippage or clinical breakage) divided by the number of condoms used during intercourse, reported as a percentage. Clinical failure events, defined in ISO 29943-1:2017, will be reported by subjects.

IPD SHARING:
Plan to Share IPD: Yes
The study information may be released to the groups listed below:
  The study sponsor (or sponsor representatives such as monitors and/or auditors) The U.S. Food and Drug Administration (FDA) Sterling Institutional Review Board (IRB) The Department of Health and Human Service (DHHS) Other government agencies in other countries Other doctors, health care professionals or research staff who are involved in the study The results of the study, including participants' information, may also be presented at meetings or in articles written about the study (publications). If the results of the study are published, the participants' identity will remain confidential.